CLINICAL TRIAL: NCT06556706
Title: Impact of Urolithin A (Mitopure) on Mitochondrial Quality in Muscle of Frail Older Adults
Acronym: MitoEM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Amazentis SA (Industry)
Collaborators: Université du Québec a Montréal (Other); McGill University Health Centre/Research Institute of the McGill University Health Centre (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: 2024-10182
Record Dates: First submitted 2024-08-09; First posted 2024-08-16 (Actual); Last update posted 2025-05-28 (Actual); Status verified 2025-05

CONDITIONS: Frailty; Sarcopenia; Aging; Muscle Atrophy
Keywords: mitophagy; Urolithin A
MeSH Terms: conditions — Frailty; Sarcopenia; Muscular Atrophy | interventions — 3,8-dihydroxy-6H-dibenzo(b,d)pyran-6-one

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Placebo (Placebo Comparator)
  Interventions: Dietary Supplement: Placebo
- Mitopure (Urolithin A) (Active Comparator)
  Interventions: Dietary Supplement: Mitopure (Urolithin A)

INTERVENTIONS:
Dietary Supplement: Mitopure (Urolithin A) — UA is produced by the gut microbiome following the digestion of dietary precursors (polyphenols such as ellagitannins and punicalagins) present in fruits and nuts such as pomegranate, nuts and berries.
  In mouse models of aging and muscle dystrophy, UA was shown to induce mitophagy and mitochondrial function in the skeletal muscle. This was associated with improved muscle strength and endurance (Nat. Med, 2016; Sci Tran Med, 2021). In humans, UA was shown to be safe and bioavailable in multiple clinical studies (Nat. Met, 2019; Cell Rep Med, 2022; JAMA Network Open, 2022).
  Arms: Mitopure (Urolithin A)
Dietary Supplement: Placebo — Placebo containing excipients other than Urolithin A (Mitopure)
  Arms: Placebo

SUMMARY:
The study is a single-center, randomized, placebo-control double-blind study in frail older adults over 65yrs. to investigate the impact of Mitopure (Urolithin A) supplementation on muscle mitochondrial quality in frail older adults after 8-weeks of supplementation

ELIGIBILITY:
Inclusion Criteria:

* Frail (as defined by the Fried frailty criteria)nonsmoking participants in the age group of 65 to 85 years old, both male and female.
* A body mass index between 18 to 35 kg/m2.
* Not on any medications/living with medical conditions that would compromise the study outcome or the safety of the research participant.
* Able to participate and willing to give written informed consent and to comply with the study restrictions.
* Willing to be assigned randomly either to the UA or the control group.

Exclusion Criteria:

Participants must not have:

* Participated in a clinical trial within 90 days of screening or more than 4 times in the previous year.
* A history (within 3 months of screening) of alcohol consumption exceeding 2 standard drinks per day on average (1 standard drink = 10 grams of alcohol).
* A history or presence of allergy to 5-aminolevulinic acid or porphyrins.
* A history or presence of allergy to lidocaine.
* Positive hepatitis B surface antigen (HBsAg), hepatitis C antibody (HCV Ab), or human immunodeficiency virus antibody (HIV Ab) at screening.
* Unwillingness or inability to refrain from consuming alcohol within 48 hours before each visit until the end of said visit.
* Unwillingness or inability to refrain from consuming 8 or more units of xanthine containing beverages and foods per day during the entire study.
* Unwillingness to not consume other mitochondrial supplements during the course of the study (such as CoQ10, reseveratrol, NR, NMN etc.) and pomegranate juice
* unwillingness to not change diet or physical activity levels during the course of the study
* Unwillingness or inability to undergo a muscle biopsy.
* Underlying chronic disease, which in the opinion of the investigator, would interfere with study participation or the validity of the measurements.
* Unintentional weight loss ≤5% of regular body weight during the last 6 months.
* Medication requirements that may interfere with the interpretation of the results.
* Loss or donation of blood over 500mL three months prior (male subjects) or four months prior (female subjects) to participating in the study.
* Smoked (tobacco and/or marijuana mixed with tobacco (THC)) within 6 months prior to the start of the study;
* Abused drugs, medicine or alcohol within up to 30 days prior to the start of the study (Alcohol: more than 10 drinks a week, with more than 2 drinks a day most days; Drugs: THC, cocaine, opiates, amphetamines/methamphetamines, benzodiazepines, barbiturates, Buprenorphine, Creatin, Methadone metabolite, oxycodone, phencyclidine);
* A positive COVID-19 test taken 1 week to 24h before study start date.

Ages: 65 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 26 (Actual)
Dates: Start 2024-08-15 (Actual); Primary Completion 2025-04-25 (Actual); Study Completion 2025-04-25 (Actual)

PRIMARY OUTCOMES:
Change in mitochondrial area between placebo and active treated groups assessed via Electron Microscopy | 8-weeks
Change in mitochondrial cristae density between placebo and active treated groups assessed via Electron Microscopy | 8-weeks

SECONDARY OUTCOMES:
change between groups on the following: maximal mitochondrial O2 consumption assessed via via respirometry on permeabilized myofibers | 8-weeks
change between groups in mitochondrial calcium retention capacity measured by mitochondrial permeability transition pore (mPTP) sensitivity to calcium | 8-weeks
mitochondrial DNA (mtDNA) over nuclear DNA ratio (mtDNA/nDNA) via qPCR | 8-weeks
Changes in body composition via Dual X-ray Absorptiometry (DXA) scan of total and appendicular lean mass | 8-weeks
Changes in composition via Peripheral quantitative computed tomography (pQCT) of muscle tissue | 8-weeks
Changes in the timed up and go test (time needed to stand from an armchair, walk a distance of 3 meters, turn around and sit back down in the chair) | 8-weeks
Changes in grip strength measured by a hand dynamometer | 8-weeks
Changes in Berg balance test: Participant will be asked to maintain a given position or perform a task | 8-weeks
Changes in distance walked during the six-minute walk test | 8-weeks
Changes in the 30-second stand test: Participant will stand as many times as s/he can from a seated position for 30-seconds. | 8-weeks
Changes in Four-square step test: To assess balance, participant will step over small sticks placed in an X on the floor | 8-weeks
Changes in Unipedal stance test (UPST): First a ball will be kicked to determine dominant leg, then participant will be asked to stand on one leg (barefoot) with eyes open and again with eyes closed | 8-weeks
Recording of adverse events | 8-weeks
Quantification of muscle fiber type (type I/II) via Myosin Heavy Chain immunolabeling | 8-weeks
Analysis of markers of neuromuscular junction integrity (NCAM biomarker staining) | 8-weeks
Changes in knee extension strength measured by a hand dynamometer | 8-weeks

CONTACTS AND LOCATIONS:
Overall Officials: José Morais, Principal Investigator — McGill University Health Centre/Research Institute of the McGill University Health Centre; Gilles Gouspillou, PhD, Principal Investigator — UQAM (University of Quebec at Montreal)
Locations (1):
- McGill University Health Center, Montreal, Canada

IPD SHARING:
Plan to Share IPD: No